CLINICAL TRIAL: NCT01530451
Title: Prospective, Randomized, Double-blind Trial of Desmopressin on Nocturia in Obstructive Sleep Apnoea Patients
Brief Title: Clinical Trial of Desmopressin on Nocturia in Obstructive Sleep Apnoea Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Eddie SY Chan, MD, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NOCOSA-001
Record Dates: First submitted 2012-02-02; First posted 2012-02-10 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Nocturia; Obstructive Sleep Apnoea
Keywords: Nocturia; Obstructive sleep Apnoea; Desmopressin
MeSH Terms: conditions — Nocturia; Sleep Apnea, Obstructive | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Drug/ Placebo (Experimental): Initial phase on Desmopressin and then cross over to placebo on the second phase
  Interventions: Drug: Desmopressin; Drug: Placebo
- B: Placebo/ Drug (Experimental): Initial phase on Placebo and then cross over to Desmopressin on the second phase
  Interventions: Drug: Desmopressin; Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin — 120mg OD
  Other Names: Minirin
Drug: Placebo — one tab OD

SUMMARY:
The purpose of the study is to evaluate the efficacy of desmopressin on symptoms of nocturia in patients with Obstructive Sleep Apnoea (OSA). The improvement of sleep quality and the quality of life will be measured.

DETAILED DESCRIPTION:
Nocturia is one of the commonest urinary symptoms in elderly and in patients with obstructive sleep apnoea (OSA). According to the International Continence Society (ICS) definition, nocturia is defined as "the complaint that the individual has to wake at night one or more times to void" . It implies a continuum beginning from what might be considered normal, to a bothersome state. Bothersome nocturia is a common and age-dependent condition. A prevalence ranging from 48.6% to 77% were reported in the literature. Pathogenesis of nocturia is multi-factorial, and has closely related to OSA. OSA patients generate negative intrathoracic pressure during sleep, this leads to increased venous return and distension of the right atrium. This leads to an increase of hormone secretion, namely Atrial Natriuretic Peptide (ANP). ANP causes increased sodium and water excretion, and inhibits the secretion of antidiuretic hormone. All of the above factors results in an increased nocturnal urine production and nocturia.

Middle-aged men with OSA always present to urology clinic with lower urinary tract symptoms with predominant nocturia. Many a time they were treated as benign prostatic hyperplasia with multiple medications with suboptimal response. The underlying genuine pathology of OSA-related nocturia is overlooked.

Desmopressin is an analogue of antidiuretic hormone, it is the pharmacological therapy of choice for patients with nocturia where night-time polyuria is present.

In this study, the investigators would like to evaluate the efficacy of desmopressin on symptoms of nocturia in patients with Obstructive Sleep Apnoea (OSA). The improvement of sleep quality and the quality of life will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patient (aged</=65 years old)
* Obstructive sleep apnoea diagnosed by sleep study
* Stable treatment on obstructive sleep apnoea and / or LUTS
* Nocturia on average more than once per night
* Having the ability to communicate and comply with the requirements of the study

Exclusion Criteria:

* Presence of urethral strictures and neurogenic bladder dysfunction
* Clinical evidence of bladder stones, bladder tumor or an active urinary tract infection
* History of prostate cancer or prostate specific antigen (PSA) level > 10ng/ml or suspicious of prostate cancer on digital rectal examination (DRE), unless a transrectal biopsy of prostate has been performed and the presence of prostate cancer has been excluded.
* Patient on intermittent self-catheterisation
* Recent start or change of treatment on obstructive sleep apnoea and / or nocturia
* Uncontrolled medical problems: e.g. Diabetes Mellitus or Diabetes insipidus
* Hyponatraemia
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in no. of nocturia | Week 4 and Week 13

SECONDARY OUTCOMES:
Side effects related to desmopressin | up to Week 13
Change in quality of Life - NQOL | Week 4 and Week 13
Change of quality of Sleep - PSQI | Week 4 and Week 13
Change in lower urinary tract symptoms - OABSS | Week 4 and Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Eddie SY Chan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong